CLINICAL TRIAL: NCT02334345
Title: Skin Protection During Radiotherapy in Patients With Breast Cancer: A Comparative Study of Evoskin® Verus Trixéra®
Brief Title: Skin Protection During Radiotherapy in Patients With Breast Cancer
Acronym: EVOSKIN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Limoges (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: I13026
Record Dates: First submitted 2014-12-16; First posted 2015-01-08 (Estimated); Last update posted 2022-03-14 (Actual); Status verified 2022-02

CONDITIONS: Radiation Dermatitis
MeSH Terms: conditions — Radiodermatitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- EVOSKIN (Experimental): Patients are to apply Evoskin ( topical agent) in the half of the irradiated breast 3 hours after radiothérapy and may be applied again later the same day.
  Interventions: Drug: Evoskin
- TRIXIERA (Active Comparator): Patients are to apply Trixiera ( topical agent) in the other half of the irradiated breast 3 hours after radiothérapy and may be applied again later the same day.
  Interventions: Drug: Trixiera

INTERVENTIONS:
Drug: Evoskin — Evoskin is Trixiera is a topical agent recommended to help patients in the management of radiation skin reactions
  Arms: EVOSKIN
Drug: Trixiera — Trixiera is a topical agent recommended to help patients in the management of radiation skin reactions
  Arms: TRIXIERA

SUMMARY:
Radiotherapy may cause severe skin changes that significantly interfere with the patient's quality of life and may reduce radiotherapy effectiveness. Many skin care instructions and various topical agents are recommended to help patients in the management of radiation skin reactions, but evidence to support the value of the topical treatments of the irradiated skin is lacking. In the present study we investigated the effects of two topical agents used as supportive care to protect skin during radiotherapy.

DETAILED DESCRIPTION:
Women with breast cancer and were to receive breast radiotherapy to 50 Gy were enrolled in a prospective randomized trial to compare the effectiveness of Evoskin®) for protecting skin compared to Trixiera. To account for individual differences in radiation each subject served as her own control, as each was to apply the experimental and control agents to the irradiated breast. Each patient was randomly assigned to use Evoskin on the half of the irradiated breast and to use the Triexiera on the other half. Dermatitis was graded weekly by means of a spectrophotometer.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old or more
* Patients with breast cancer for which a treatment by radiotherapy is planned
* No concomitant chemotherapy
* Signed informed consent

Exclusion Criteria:

* Cutaneous neoplasia radiotherapy
* Total mastectomy
* Bilateral breast cancer
* Dark skinDiseases enhancing radiosensitivity Patient with a generalized skin disorder
* Pregnant, breast-feeding woman

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2015-01; Primary Completion 2015-11-01 (Actual); Study Completion 2021-01-17 (Actual)

PRIMARY OUTCOMES:
Average of the radiation dermatitis intensity | at 3 months
  Radiation dermatitis will be assessed by means of a spectrophotometer after the patient has received 50Gy

SECONDARY OUTCOMES:
Clinical grade of dermatitis | at 3 months
  dermatitis grade will be assessed according to CTCAE after the patient has received 50 Gy

CONTACTS AND LOCATIONS:
Overall Officials: Pierre CLAVRE, MD, Principal Investigator — CHU LIMOGES
Locations (1):
- CHU LIMOGES - Radiothérapie, Limoges, France